CLINICAL TRIAL: NCT02004041
Title: A Randomized, Double-Blind, Placebo-Controlled, Proof of Concept, Antipruritic Study of the Neurokinin-1 Receptor Antagonist VLY-686 in Subjects With Treatment-Resistant Pruritus Associated With Atopic Dermatitis
Brief Title: Proof of Concept of VLY-686 in Subjects With Treatment-Resistant Pruritus Associated With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VLY-686-2101; 2013-002931-25 (EudraCT Number)
Record Dates: First submitted 2013-11-21; First posted 2013-12-06 (Estimated); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Treatment-resistant Pruritus Associated With Atopic Dermatitis
Keywords: pruritus; atopic dermatitis; VLY-686
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic | interventions — LY686017

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VLY-686 (Experimental)
  Interventions: Drug: VLY-686
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VLY-686
  Arms: VLY-686
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is randomized, double-blind, placebo-controlled study to test whether VLY-686 can reduce chronic pruritus in subjects with treatment-resistant pruritus associated with atopic dermatitis in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 - 65 years, inclusive; suffering from atopic dermatitis with a SCORAD index at inclusion ≤80; with atopic lesions on arms, legs, trunk and neck;
* Chronic pruritus with pruritus being actively present for at least 6 weeks prior to screening;
* Males, non-fecund females, or females of child-bearing potential using 2 independent highly effective barrier methods of birth control when used correctly for a period of 35 days before the first dosing, during the study and for one month after the last dose and must have a negative pregnancy test at the screening and baseline visits.

Exclusion Criteria:

* Chronic pruritus due to conditions other than atopic dermatitis (AD) including the following conditions: Prurigo nodularis, Lichen simplex chronicus, Bullous pemphigoid;
* Acute superinfection of AD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2015-02-19 (Actual); Study Completion 2015-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Vanda Investigational Site, Düsseldorf
  - Vanda Investigational Site, Hamburg
  - Vanda Investigational Site, Jena
  - Vanda Investigational Site, Kiel
  - Vanda Investigational Site, Münster

RESULTS

PARTICIPANT FLOW:
Groups:
- VLY-686: VLY-686
- Placebo: Placebo
Period: Overall Study
Arm/Group | VLY-686 | Placebo
Started | 34 | 35
Completed | 30 | 31
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VLY-686 | Placebo | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (15.6) | 40.2 (14.5) | 38.4 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  Germany | 34 | 35 | 69
Pruritus 24 hours average intensity Visual Analogue Scale (VAS) at baseline [Mean (Standard Deviation); unit: units on a scale] — Responses were measured on a 100-mm Visual Analogue Scale (VAS), where the left end point was marked "no itch" (0 mm) and in the right end point was marked "worst imaginable itch" (100 mm).
  units on a scale | 76.1 (9.74) | 77.2 (10.87) | 76.6 (10.27)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint (Day 28 or Early Termination) in Visual Analogue Scale (VAS) Pruritus 24 Hour Average Intensity.
Description: Responses were measured on a 100-mm Visual Analogue Scale (VAS), where the left end point was marked "no itch" (0 mm) and in the right end point was marked "worst imaginable itch" (100 mm).
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | VLY-686 | Placebo
Number analyzed (Participants) | 34 | 33
mm | -40.5 (5.30) | -36.5 (4.96)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent through study completion (approximately 63 days) regardless of seriousness or relationship to investigational product.
Arm/Group | VLY-686 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 12/34 | 11/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VLY-686 (N=34) | Placebo (N=34)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other